CLINICAL TRIAL: NCT01075022
Title: Effect of a Single Colecalciferol Dose on Insulin Resistance: A Prospective Randomized Trial
Brief Title: Effect of a Single Colecalciferol Dose on Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Gustavo Faulhaber, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 33598290
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Insulin Resistance; Glucose Intolerance
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Drug: Colecalciferol (Vitamin D3) 300.000 UI
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colecalciferol (Vitamin D3) 300.000 UI — Colecalciferol (Vitamin D3) 300.000 UI Capsule, Single Dose
  Arms: Vitamin D
Drug: Placebo — Placebo Capsule, Single Dose
  Arms: Placebo

SUMMARY:
A Prospective Double-Blinded, Placebo Controlled, Randomized Trial comparing a single dose of Vitamin D (Colecalciferol) 300.00UI to placebo on patients with insulin resistance. Primary Outcome: Blood glucose and homeostasis model assessment for insulin resistance (HOMA-R) after 90 days. Study hypothesis: Vitamin D treatment may improve insulin resistance and decrease glucose level, since there is an association between hypovitaminosis D and increased insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Fasten Blood Glucose > 100 mg/dL and < 126 mg/dL
* Age > 18 years

Exclusion Criteria:

* Diabetes Mellitus
* Use of metformin
* Vitamin D Use
* Hypercalcemia
* Chronic Hepatitis
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Level | Baseline and day 90

SECONDARY OUTCOMES:
Blood Calcium Level | Baseline and day 90
HOMA-R | Baseline and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Tania Furlanetto, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil